CLINICAL TRIAL: NCT05186103
Title: Participation of Children With Autism Using Parental Reporting Tools Combined With a Performance-based Tool, the Washing Hands Structured Observation (WashHO).
Brief Title: Activities of Daily Living Participation Characteristics Among School-Aged Children With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Sara Rosenblum (Other)
Responsible Party: Sponsor-Investigator, Sara Rosenblum, Professor in the Department of Occupational Therapy, Faculty of Social Welfare Affiliation: University of Haifa Collaborators:, University of Haifa
Organization: University of Haifa (Other)
Other Study IDs: ADL
Record Dates: First submitted 2021-11-29; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; self care; ADL; daily function; executive functions
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HS-ASD: high-severity ASD
  Interventions: Other: observation
- LS-ASD: low-severity ASD
  Interventions: Other: observation
- control: typical development
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — The assessment combined a parent-reported questionnaire (the Participation in Childhood Occupation; PICO) alongside the Pediatric Evaluation of Disability Inventory (PEDI self-care) and a Performance-based task, the Washing Hands Structured Observation (WashHO).

SUMMARY:
This study aimed to investigate the performance of activities of daily living (ADL) among 53 children ages 6-10 years: 17 with high-severity ASD (HS-ASD), 16 with low-severity ASD (LS-ASD), and 20 controls with typical development. Methods: The assessment combined a parent-reported questionnaire (the Participation in Childhood Occupation; PICO) alongside the Pediatric Evaluation of Disability Inventory (PEDI self-care) and Performance-based task, the Washing Hands Structured Observation (WashHO).

DETAILED DESCRIPTION:
study objectives were to:

(a) Examine participation characteristics in self-care and daily activities of school-age children with HS-ASD and LS-ASD compared to children with typical development, based on the parent-reported Participation in Childhood Occupation Questionnaire (PICO-Q) for ASD and PEDI (b) Establish the validity and reliability of the WashHO assessment.

The research hypotheses were (A) Significant differences will be found among children with HS-ASD, children with LS-ASD, and children with typical development in results of the PICO-Q and the PEDI self-care subtest of independence.

(B1) The internal consistency of the WashHO assessment will be at a Cronbach alpha level equal to or greater than 70.

(B2) Significant differences will be found among children with HS-ASD, LS-ASD, and typical development in the WashHO assessment performance criteria, thus establishing the WashHO's discriminate validity.

(B3) Significant correlations will be found among the four PICO-Q ADL items, which involve performing a sequence of actions (bathing, hygiene, clothing, and washing hands) and the WashHO assessment performance scores, establishing its convergent validity.

(B4) Significant correlations will be found among the WashHO performance and degree of independence scores and the PEDI independence subtest in self-care, establishing the WashHO's concurrent validity.

ELIGIBILITY:
Inclusion Criteria:

Hebrew speakers

* study groups- ASD diagnosis provided by pediatricians or clinical psychologists according to DSM-5 criteria (APA, 2013).

Exclusion Criteria:

* without ASD formal diagnosis

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study participants with an ASD diagnosis were recruited from special education schools, special education classes located in regular schools, or mainstream schools through parent referral.no significant group differences were found for the participants' age, gender, socioeconomic status, or religion.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
PICO-Q ASD | through study completion, an average of 3 Months
  The 34-item PICO-Q for ASD measures the level, enjoyment, and frequency of performance for children's participation in daily occupations in five domains: ADL (16 items), academic activity (seven items), play and leisure (four items), social functioning (four items), and routines and habits (two items; Bar-Shalita et al., 2009; Heller., 2013). In this study, each child could choose two addition items in which they were participating, and a handwashing item was added. Each item has four scores: difficulty in performance, frequency, involvement, and level of enjoyment, and scores range from 1 (low) to 5 (high).
PEDI Self-Care Subtest | through study completion, an average of 3 Months
  Pediatric Evaluation of Disability Inventory- parent report about children's ADL performance abilities (Haley et al., 1992). The test includes eight items measuring the typical amount of assistance the caregiver provides during the child's completion of tasks such as eating, grooming, and handwashing. Each item is scored from 5 (independence, no physical assistance or supervision) to 0 (total assistance, the caregiver does the entire task) and includes scoring of frequency-type adjustments. The total scale score ranges between 0 and 100, with lower scores indicating higher severity levels.
the Washing Hands Structured Observation (WashHO) | through study completion, an average of 3 Months
  was developed based on the Do-Eat Performance-Based Assessment for Children (Do-Eat; Josman et al., 2010). examines BADL performance, sensorimotor skills, and executive functions abilities across the child's natural environments. includes four domains (a) performance analysis (10 items), (b) sensorimotor skills (SM; six items), (c) executive functions (EF; nine items), and (d) 10 unique performance characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Rosenblum, Phd, Study Director — University of Haifa
Locations (1):
- Hana Levy-Dayan, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided